CLINICAL TRIAL: NCT04242485
Title: Osteopathy Treatment Restores Cardiovascular Autonomic Parameters in Rugby Players
Brief Title: Osteopathy Treatment and Cardiovascular Recovery After a Rugby Match
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: Collegio Italiano di Osteopatia (Unknown); Foundation COME Collaboration (Unknown)
Responsible Party: Principal Investigator, Elena Giovanna Bignami, full professor, University of Parma
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 032017
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cardiovascular Physiological Phenomena
Keywords: heart rate; heart rate variability; blood pressure; rugby match; atlethes; recovery; osteopathy
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AFTER MATCH + OMT (Other): Players undertook a recording session the day after a rugby match and received osteopathic manipulative treatment
  Interventions: Other: Osteopathic manipulative treatment
- AFTER MATCH + sham treatment (Other): Players undertook a recording session the day after a rugby match and received sham treatment
  Interventions: Other: Sham treatment
- NO MATCH + OMT (Other): Players undertook a recording session the day after a resting day and received osteopathic manipulative treatment
  Interventions: Other: Osteopathic manipulative treatment
- NO MATCH + sham treatment (Other): Players undertook a recording session the day after a resting day and received sham treatment
  Interventions: Other: Sham treatment

INTERVENTIONS:
Other: Osteopathic manipulative treatment — Each osteopathic manipulative treatment consisted of a structured evaluation to diagnose somatic dysfunction of the pelvis, abdomen, vertebral spine, and upper and lower limbs (10 min), followed by the therapeutic application of manually guided forces to improve physiological function and homeostasis that has been altered by somatic dysfunction for 20 min, using techniques that were left at the discretion of the osteopath, including the myofascial release and cranial sacrum techniques
  Arms: AFTER MATCH + OMT; NO MATCH + OMT
Other: Sham treatment — The sham treatment consisted only in "soft touch" of the same body areas involved in the osteopathic manipulative treatment protocol without applying any pressure
  Arms: AFTER MATCH + sham treatment; NO MATCH + sham treatment

SUMMARY:
The purpose of this study was to explore the efficacy of osteopathic manipulative treatment (OMT), a form of non-invasive manual treatment, for a faster recovery of cardiovascular parameters after a rugby union match in professional male athletes. To this end, the effects of OMT on resting cardiovascular function and cardiovascular reactivity were evaluated in twenty-three male players 18-20 hours after a match and compared with a corresponding no-match (control) condition. Assessment of resting cardiovascular parameters 18-20 hours after a match revealed the presence of elevated mean arterial pressure and heart rate, and reduced vagally-mediated heart rate variability compared with a no-match condition. OMT provoked a significant reduction in mean arterial pressure and increased vagally-mediated heart rate variability at rest both in the after match and control conditions. Moreover, OMT favoured a larger vagal withdrawal in response to an orthostatic stress compared with a sham treatment. These results suggest that OMT may be implemented as a recovery strategy to restore athletes' cardiovascular homeostasis after a rugby union match.

DETAILED DESCRIPTION:
The presence of cardiovascular autonomic alterations in the aftermath of an intense exercise performed during a competitive match may indicate incomplete recovery and prolonged fatigue.Therefore, the implementation of effective interventions aimed at favoring a faster recovery of athletes' cardiovascular homeostasis in the aftermath of a competitive match may be beneficial for greater adaptations to subsequent training and enhanced overall performance. In this regard, osteopathic manipulative treatment (OMT) is a form of non-invasive manual treatment that uses a set of touch, manipulation and mobilization procedures to diagnose, treat, and prevent illness or injury. In the present study, the investigators sought to explore the efficacy of a single session of OMT in restoring alterations in cardiovascular parameters at rest and in response to an orthostatic challenge in trained adult male athletes long after (18-20 hours) a rugby union match.

ELIGIBILITY:
Inclusion Criteria:

* being healthy and injury-free
* age ≥ 18 years old
* being Caucasian
* regular participation in competitive matches of rugby union consisting of 2, 40-min halves
* regular training for an average of six hours/week during the last four weeks

Exclusion Criteria:

* history of cardiovascular disease or traumatic brain injury
* chronic drug treatment
* use of any medications during the last week
* having received osteopathic manipulative treatment before

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Resting heart rate | ECG recorded for 10 min just before osteopathic manipulative treatment and sham treatment
  Mean heart rate measured as beats per minute
Resting heart rate | ECG recorded for 5 min just after osteopathic manipulative treatment and sham treatment
  Mean heart rate measured as beats per minute
Resting heart rate variability (RMSSD index) | ECG recorded for 10 min just before osteopathic manipulative treatment and sham treatment
  Root mean square of the successive differences between adjacent heart beats (RMSSD) measured in ms
Resting heart rate variability (RMSSD index) | ECG recorded for 5 min just after osteopathic manipulative treatment and sham treatment
  Root mean square of the successive differences between adjacent heart beats (RMSSD) measured in ms
Resting heart rate variability (HF index) | ECG recorded for 10 min just before osteopathic manipulative treatment and sham treatment
  High frequency (HF) component power of the RR interval spectrum measured in ms2
Resting heart rate variability (HF index) | ECG recorded for 5 min just after osteopathic manipulative treatment and sham treatment
  High frequency (HF) component power of the RR interval spectrum measured in ms2
Resting mean arterial pressure | Assessed just before osteopathic manipulative treatment and sham treatment with a sphygmomanometer
  Mean arterial pressure measured in mmHg
Resting mean arterial pressure | Assessed just after osteopathic manipulative treatment and sham treatment with a sphygmomanometer
  Mean arterial pressure measured in mmHg

SECONDARY OUTCOMES:
Heart rate reactivity to orthostasis | ECG recorded for 10 min during orthostasis (5 min) and subsequent recovery (5 min)
  Mean heart rate measured as beats per minute
Heart rate variability (RMSSD index) reactivity to orthostasis | ECG recorded for 10 min during orthostasis (5 min) and subsequent recovery (5 min)
  Root mean square of the successive differences between adjacent heart beats measured in ms
Heart rate variability (HF index) reactivity to orthostasis | ECG recorded for 10 min during orthostasis (5 min) and subsequent recovery (5 min)
  High frequency component power of the RR interval spectrum measured in ms2

CONTACTS AND LOCATIONS:
Locations (1):
- Collegio Italiano di Osteopatia, Parma, Italy

IPD SHARING:
Plan to Share IPD: No